CLINICAL TRIAL: NCT02951585
Title: Pilot, Prospective, Comparative Multicentric Study Evaluating the Effects on the Arthrosis Biomarkers, the Clinical Effectiveness, the Tolerance of an Intra-articular Injection of Hyaluronic Acid KARTILAGE CROSS Versus Placebo in Patients Suffering From Knee Osteoarthritis.
Acronym: EPIKART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Vivacy (Industry)
Collaborators: Artialis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-A01521-42
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- KARTILAGE CROSS (Experimental): Kartilage® Cross (2.2 mL, 16 mg/g of hyaluronic acid)
  Interventions: Device: KARTILAGE CROSS
- Placebo (Placebo Comparator): Saline solution (2.2-2.5 mL, NaCl 9 mg/g)
  Interventions: Device: PLACEBO

INTERVENTIONS:
Device: KARTILAGE CROSS — Intra-articular injection of Kartilage Cross
  Arms: KARTILAGE CROSS
Device: PLACEBO — Intra-articular injection of physiological serum (saline solution)
  Arms: Placebo

SUMMARY:
Intra-articular hyaluronic acid injections, also known as viscosupplementation, are a treatment option for knee osteoarthritis that serves to restore the decreasing rheological properties of synovial fluid. KARTILAGE® CROSS is a visco-elastic gel of highly purified reticulated hyaluronic acid. It contains mannitol to provide an anti-oxidative action and to avoid hyaluronic acid depolymerization. Reticulation and mannitol increase the residency time of the product in the joint cavity then allowing a single injection in painful knee osteoarthritis patients.

The US food and drugs administration (FDA) and European medicine agency (EMA), have recently published guidelines recommending a higher level of integration of biomarkers in the development and testing of new drugs to advance decision-making on dosing, time and treatment effect, trial design, and risk/benefit analysis. Biomarkers can be used not only in the process of drug development, but also in the future in assessment of individual patient's response to treatment.

Several soluble biomarkers have been identified as potential candidates to predict or monitor the efficacy of intervention. Coll2-1, a degradation product of type II collagen, and Coll2-1NO2, a nitrated form of the Coll2-1 peptide have been studied in human osteoarthritis and entered the qualification process. Evidences demonstrated them to be pertinent and to be foresee as markers used for the diagnosis, the prognosis, the burden of disease and the monitoring of a treatment efficacy.

The aim of this study was to provide with the first kinetic data regarding biomarkers in painful knee osteoarthritis patients treated with a new reticulated hyaluronic acid. The effects of the treatment were compared to those of saline solution. The primary endpoint was a specific osteoarthritis biomarker, Coll2-1. The secondary endpoints were the effects of the treatment or placebo on other biomarkers of osteoarthritis, its clinical efficacy and tolerance

ELIGIBILITY:
Inclusion Criteria:

* Man or Women, aged from 45 to 80
* Presenting a symptomatic femoro-tibial knee osteoarthritis responding to clinical and radiologic ACR (American College of Rheumatology) criteria,
* Symptomatic since at least 6 months
* Mean global knee pain determined on Visual Analog Scale for the last 24 hours over 40 mm (without any NSAIDs or analgesics for more than 48 hours).
* Kellgren and Lawrence (K&L) radiological stage must have been II or III on pictures lasted less than 12 months
* Requiring a treatment with hyaluronic acid after failure or intolerance to first line analgesics or NSAIDs
* Having signed an informed consent after receiving comprehensive information
* Capable to follow the study instructions
* Benefiting from health insurance.

Exclusion Criteria:

Related to the osteoarthritis pathology:

* Significant clinical knee effusion
* Radiographical Kellgren and Lawrence grade I or IV
* Osteoarthritis secondary to a microcrystalline arthropathy: chondrocalcinosis previously known or defined by a calcium border on at least one tibiofemoral spacing, gout ...
* Isolated femoropatellar osteoarthritis
* Presence of another joint (other than the evaluated knee) affected by osteoarthritis (known and symptomatic): collateral knee, hip, hand, shoulder, ankle or foot
* Chondromatosis or villonodular synovitis of the knee
* Paget disease
* Recent trauma (< 1 month) of the evaluated knee
* Pathologies interfering with the evaluation of osteoarthritis (microcrystalline inflammatory arthropathy, rheumatoid arthritis, radiculalgia in the lower limbs, arteritis. etc)
* Acute inflammatory osteoarthritis (Kofus ≥ 7)

Related to previous and concomitant treatments

* Corticosteroids injection in the last month before injection regardless the concerned joint
* Hyaluronan injection in the last 6 months before injection regardless the concerned joint
* Analgesics and NSAIDs intake during the last 48 hours before inclusion visit
* Change in the dosage of slow-acting drugs against arthrosis i.e. chondroitin, glucosamine, diacerein or avocado-soybean unsaponifiables in the last 3 months before inclusion or planned during study
* Arthroscopy or surgery in the target knee in the last 3 months before inclusion
* Oral corticotherapy

Related to associated pathologies

* Severe diseases (severe hepatic failure, renal failure, uncontrolled cardiovascular diseases….)
* Dermatological infection at the site of injection
* Anticoagulant treatment
* Risk of hemorrhage according to the evaluator or injector assessment

Related to the patients

* Known allergy to hyaluronan
* Known allergy to acetaminophen
* Known allergy to mannitol
* Pregnant or breastfeeding women
* Premenopausal women without contraception
* Patient unable to read, and to write
* Patient having participated in a clinical research investigation in the last 3 months
* Patient under guardianship or judicial protection

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patient with a reduction of at least 10 nmol/l of serum Coll2-1 between inclusion visit (10 days before injection) and 3 months after injection. | 3 months after injection

SECONDARY OUTCOMES:
Variation in Coll2-1 between inclusion and 1 month or 6 months; | 1 month and 6 months
Variation of Lequesne index (LI) between inclusion visit and further visits | 1 month, 3 months and 6 months
Variation in the global assessment of pain with visual analog scale (0-100 mm) between inclusion visit and further visits, | 1 month, 3 months and 6 months
Percentage of responders according to OMERACT/OARSI (Outcome Measures in Rheumatoid Arthritis Clinical Trials/Osteoarthritis Research Society International) at 3 months and 6 months | 3 months and 6 months
Acetaminophen and Nonsteroidal anti-inflammatory drugs (NSAID) consumption during the study | 1 month, 3 months and 6 months
Patient's global assessment of the disease activity | 1 month, 3 months and 6 months
Monitoring of adverse events | 1 month, 3 months and 6 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henrotin Y, Berenbaum F, Chevalier X, Marty M, Richette P, Rannou F. Reduction of the Serum Levels of a Specific Biomarker of Cartilage Degradation (Coll2-1) by Hyaluronic Acid (KARTILAGE(R) CROSS) Compared to Placebo in Painful Knee Osteoarthritis Patients: the EPIKART Study, a Pilot Prospective Comparative Randomized Double Blind Trial. BMC Musculoskelet Disord. 2017 May 26;18(1):222. doi: 10.1186/s12891-017-1585-2. PMID 28549430